CLINICAL TRIAL: NCT03122756
Title: Effect of Intravenous Dexamethasone Before Spinal Anesthesia on Post-cesarean Section Pain: Randomized Controlled Trial
Brief Title: Effect of Intravenous Dexamethasone Before Spinal Anesthesia on Post-cesarean Section Pain
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Principal Investigator, Abdelhameed Ahmed Ali Ismail, Dr, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IVD-SA-CS
Record Dates: First submitted 2017-04-12; First posted 2017-04-21 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Cesarean Section
Keywords: Intravenous Dexamethasone; Spinal Anesthesia; Post-cesarean Section Pain
MeSH Terms: interventions — Dexamethasone; Calcium Dobesilate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group (D) (Experimental): will include 50 women who will receive intravenous dexamethasone.
  Interventions: Drug: Dexamethasone
- Group (C) (Placebo Comparator): will include 50 women who will receive intravenous normal saline (0.9 %).
  Interventions: Other: Normal Saline

INTERVENTIONS:
Drug: Dexamethasone — Intravenous injection of dexamethasone 0.1 mg/kg maximum 8 mg (diluted with distilled water to 2 mL) just prior to administration of spinal anesthesia.
  Other Names: Decadron
  Arms: Group (D)
Other: Normal Saline — Intravenous injection 2 mL intravenous normal saline (0.9 %) just prior to administration of spinal anesthesia.
  Arms: Group (C)

SUMMARY:
*Aim of the Work This study aims to assess the efficacy of intravenous injection of dexamethasone prior to spinal anesthesia in reducing post-cesarean section pain in women undergoing cesarean section.

DETAILED DESCRIPTION:
*Research Hypothesis: In women undergoing cesarean section, intravenous injection of dexamethasone prior to spinal anesthesia may reduce post-cesarean section pain.

*Research Question: In women undergoing cesarean section, does injecting intravenous dexamethasone prior to spinal anesthesia reduce post-cesarean section pain?

ELIGIBILITY:
* Inclusion Criteria:

  * A gestational age of 38 weeks or more and planned for elective cesarean section.
  * Living fetus.
  * Any number of previous cesarean section.
  * Intact amniotic membranes.
  * No history of bleeding tendency.
* Exclusion Criteria:

  * Refuse to participate after counseling.
  * Contraindication to spinal anesthesia (coagulopathy significant hypovolemia systemic or local sepsis - increased intracranial pressure - local anesthetic or fentanyl allergy).
  * High risk pregnancies as pre-eclampsia, any medical disorder (diabetes mellitus, cardiac disease or and thyroid disease).
  * Contraindication to corticosteroids e.g. systemic fungal infection
  * Steroid medication one week before the operation.
  * Chronic pain or daily intake of analgesic.
  * Abnormal placentation e.g. placenta previa.
  * Intrauterine infection.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women who will be planned for elective cesarean section.
Enrollment: 100 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
change in post-cesarean pain | 2, 4, 8 and 12 hours after the procedure
  post-cesarean pain degree scored by the patient on Visual Analogue Scale

SECONDARY OUTCOMES:
sensory recovery | 2, 4, 8 and 12 hours after the procedure
  sensory recovery time by cold object
motor recovery | 2, 4, 8 and 12 hours after the procedure
  motor recovery time on Bromage scale
nausea | 2, 4, 8 and 12 hours after the procedure
  postoperative nausea
vomiting | 2, 4, 8 and 12 hours after the procedure
  postoperative vomiting
shivering | 2, 4, 8 and 12 hours after the procedure
  postoperative shivering

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud AA ElShourbagy, MD, Study Chair — Professor of Obstetrics and Gynecology; Dalia A Nasr, MD, Study Director — Professor of Anesthesia, Intensive Care and Pain; Bassem A Islam, MD, Study Director — Lecturer in Obstetrics & Gynecology; Abdelhameed AA Ismail, MBBCh, Principal Investigator — Resident of Obstetrics & Gynecology
Locations (1):
- Ain Shams Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No